CLINICAL TRIAL: NCT06484972
Title: A Multicenter Cluster Randomized Controlled Study to Evaluate Guideline Adoption Through Lung Cancer Clinical Care Quality Improvement Project (QIP) in Pulmonary and Critical Care Medicine (PCCM) Department
Brief Title: A Study to Evaluate Guideline Adoption Through Quality Improvement Project (QIP) in Pulmonary and Critical Care Medicine (PCCM) Department
Acronym: LC PCCM QIP
Status: Not yet recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Wang Chen, Director of the National Center for Respiratory Medicine, China-Japan Friendship Hospital
Other Study IDs: ESR-24-22776
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Quality improvement project arm: The Quality improvement project(QIP) arm will perform QIP intervention. Patients in the QIP arm will be enrolled after about 3-month QIP intervention. The QIP interventions include: establish a coaching committee, quality improvement workshop, implementation of quality improvement measures, as well as evaluation periodically and feedback.
- Control arm: The control arm will not receive intervention and continue with usual care.

SUMMARY:
This is a cluster randomized controlled trial with PCCM department in each site being the cluster. Fifty-four sites' PCCM departments will be randomized to the QIP arm versus control arm in 2:1 allocation ratio. The QIP arm will perform QIP intervention. The control arm will not receive intervention and continue with usual care.

The primary endpoints of this study are molecular testing rate of non-small cell lung cancer (NSCLC) prior to the first systematic anti-tumor therapy, and adjuvant or first line targeted therapy treatment rate in actionable oncogenic alterations (AGA) NSCLC.

DETAILED DESCRIPTION:
Approximately 1728 patients from 54 sites will be enrolled (about 30 NSCLC [20%-30% squamous cases] and 2 extensive-stage small-cell lung cancer [ES-SCLC] patients in each site). Patients in the QIP arm will be enrolled after about 3-month QIP intervention. Patients in the control arm will be enrolled as soon as the trial starts. Data on lung cancer diagnosis and treatment pattern will be collected.

ELIGIBILITY:
1. Cluster 1.1 Cluster inclusion criteria 1.1.1 PCCM department in Tier 3 hospital. 1.1.2 PCCM department's standardized construction certification is "qualified ".

   1.1.3 PCCM department who want to improve lung cancer healthcare quality and agree to participate in study.

   1.2 Cluster exclusion criteria 1.2.1 PCCM department does not carry out anti-tumor treatment for lung cancer. 1.2.2 PCCM department participant in other lung cancer quality improvement study.
2. Individual Patient 2.1 Individual inclusion criteria 2.1.1 Pathology diagnosed NSCLC or ES-SCLC. 2.1.2 No prior systematic anti-tumor therapy, or prior adjuvant and neo-adjuvant therapies, definitive radiation/chemoradiation are permitted as long as treatment was completed at least 12 months prior to the development of recurrent disease.

2.1.3 Performance score (PS) 0-2. 2.1.4 Life expectancy >12 weeks. 2.2 Individual exclusion criteria 2.2.1 Have a plan to transfer to other hospitals to receive anti-tumor therapy within 3 months after signing the ICF.

2.2.2 Participating in another interventional clinical study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pulmonologists in PCCM(Pulmonary and Critical Care Medicine).
Sampling Method: Probability Sample
Enrollment: 1728 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Molecular testing rate of NSCLC(Non-small cell lung cancer) prior to the first systematic anti-tumor therapy | Baseline, 3/6/12/21/30 months post enrollment
  The percentage of patients with a pathological diagnosis of NSCLC who undertake molecular testing prior to the first systematic anti-tumor therapy in patients with a pathological diagnosis of NSCLC.
Adjuvant or first line targeted therapy treatment rate in AGA(Actionable oncogenic alterations) NSCLC(Non-small cell lung cancer) | Baseline, 3/6/12/21/30 months post enrollment
  The percentage of patients with AGA NSCLC who receive adjuvant or first line targeted therapy in patients with AGA NSCLC who receive adjuvant or first line systematic therapy.

SECONDARY OUTCOMES:
TNM stage diagnosis rate prior to the first anti-tumor therapy | Baseline
  The percentage of patients with clinical TNM staging diagnosis before first anti-tumor treatment of lung cancer in patients with first anti-tumor treatment of lung cancer.
Biopsy method | Baseline, 3/6/12/21/30 months post enrollment
  Describe the pathological biopsy method of lung cancer patients, including but not limited to bronchoscopy biopsy rate, percutaneous lung biopsy rate, thoracoscopic lung biopsy rate, etc.
Spirometry rate | Baseline
  The percentage of patients with lung cancer who perform spirometry in patients with lung cancer.
First line immunotherapy treatment rate in unresectable non-AGA(Actionable oncogenic alterations) NSCLC(Non-small cell lung cancer) | Baseline, 3/6/12/21/30 months post enrollment
  The percentage of patients with unresectable non-AGA NSCLC who receive first line immunotherapy in patients with unresectable non-AGA NSCLC who receive the first systematic therapy.
First line chemotherapy-immunotherapy treatment rate of ES-SCLC(Extensive-stage small-cell lung cancer) (stage III-IV) | Baseline, 3/6/12/21/30 months post enrollment
  The percentage of patients with ES-SCLC (stage III-IV) who receive first line chemotherapy-immunotherapy in patients with ES-SCLC (stage III-IV) who receive the first systematic therapy.
Surgical rate of stage I-IIIA NSCLC(Non-small cell lung cancer) | Baseline, 3/6/12/21/30 months post enrollment
  The percentage of patients with stage I-IIIA NSCLC who undergo surgical resection in patients with stage I-IIIA NSCLC.
MDT(Multi-disciplinary team) rate of stage IIIB-IV NSCLC(Non-small cell lung cancer) | Baseline, 3/6/12/21/30 months post enrollment
  The percentage of patients with stage IIIB-IV NSCLC discussed at the MDT meeting in patients with stage IIIB-IV NSCLC.
ORR(Objective response rate) of stage IIIB-IV NSCLC(Non-small cell lung cancer) | Baseline, 3/6/12/21/30 months post enrollment
  ORR will be defined as the proportion of patients who achieved BOR of a CR or PR assessed by pulmonologists.
ORR(Objective response rate) of ES-SCLC(Extensive-stage small-cell lung cancer) | Baseline, 3/6/12/21/30 months post enrollment
  ORR will be defined as the proportion of patients who achieved BOR of a CR or PR assessed by pulmonologists.
PFS(Progression-free survival) of stage IIIB-IV NSCLC(Non-small cell lung cancer) | Baseline, 3/6/12/21/30 months post enrollment
  PFS will be defined as the time from beginning of first-line treatment to disease progression or death for any cause, whichever occurs first.
PFS(Progression-free survival) of ES-SCLC(Extensive-stage small-cell lung cancer) | Baseline, 3/6/12/21/30 months post enrollment
  PFS will be defined as the time from beginning of first-line treatment to disease progression or death for any cause, whichever occurs first.
DFS(Disease free survival) of NSCLC(Non-small cell lung cancer) who receive neoadjuvant/adjuvant therapy | Baseline, 3/6/12/21/30 months post enrollment
  DFS will be defined as the time from surgery to recurrence of tumor or death for any cause, whichever occurs first.

IPD SHARING:
Plan to Share IPD: No